CLINICAL TRIAL: NCT04482647
Title: Breathing Techniques and Meditation for Health Care Workers During COVID-19
Brief Title: Breathing Techniques and Meditation for Health Care Workers During COVID-19 Pandemic
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0483; NCI-2020-04931 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0483 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-07-21; First posted 2020-07-22 (Actual); Results first posted 2022-02-16 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19 | interventions — Meditation; Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (video, breathing techniques, meditation) (Experimental): Patients view an instructional video on breathing techniques and meditation. Patients then perform breathing techniques over 3 minutes and meditation over 2 minutes BID for 28 days.
  Interventions: Other: Media Intervention; Procedure: Meditation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Yoga

INTERVENTIONS:
Other: Media Intervention — View instructional video
Procedure: Meditation Therapy — Perform meditation
  Other Names: Meditation
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Yoga — Perform breathing techniques
  Other Names: Yoga Therapy

SUMMARY:
This phase I trial investigates breathing techniques and meditation for health care workers during COVID-19 pandemic. Breathing techniques and medication may help manage stress and improve lung health. The goal of this trial is to learn if breathing techniques and meditation may help to reduce stress and improve lung health in health care workers during the COVID-19 pandemic.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate the feasibility of a short pranayama or breathing techniques and meditation during Covid-19 pandemic.

SECONDARY OBJECTIVES:

I. To determine the adherence to the practice assessed as at least 50% of participants implement the intervention for 3 or more times in a week by the end of week 1/day 7 (+ 3 days).

II. To determine the change in resilience, perceived stress and psychological impact from day 0 today 28 as measured by the Brief Resilient Coping Scale (BRCS), Perceived Stress Scale (PSS4), and COVID-19 Stress among health care workers questionnaire.

III. To determine the changes in breath holding time measured weekly for 4 weeks.

IV. To determine the differences in breath holding time between those who are adherent and those who are not adherent to the practice.

OUTLINE:

Patients view an instructional video on breathing techniques and meditation. Patients then perform breathing techniques over 3 minutes and meditation over 2 minutes twice daily (BID) for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to read and understand English
* Must be employed at MD Anderson Cancer Center

Exclusion Criteria:

* Epilepsy
* Brain tumor
* Brain aneurysm
* Pregnant or trying to get pregnant
* Brain bleeding in the past 1 year
* Recent abdominal surgery and not cleared to exercise

Max Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2027-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Santhosshi Narayanan, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Wagner RW, Mallaiah S, Anderson CR, Engle R, Vasu V, Bruera E, Subramaniam B, Cohen L, Narayanan S. Effects of the Brief Simha Kriya Breathing Practice for Health Care Workers During the COVID-19 Pandemic. J Integr Complement Med. 2024 Oct;30(10):970-977. doi: 10.1089/jicm.2023.0692. Epub 2024 Mar 28. PMID 38546421
- [Derived] Narayanan S, Tennison J, Cohen L, Urso C, Subramaniam B, Bruera E. Yoga-Based Breathing Techniques for Health Care Workers During COVID-19 Pandemic: Interests, Feasibility, and Acceptance. J Altern Complement Med. 2021 Aug;27(8):706-709. doi: 10.1089/acm.2020.0536. Epub 2021 Apr 9. PMID 33835830

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The purpose of this study is to determine the effects of web-based breathing techniques and meditation on lung health and building resilience among health care workers dealing with the COVID-19 pandemic.
Period: Overall Study
Arm/Group | Supportive Care (Video, Breathing Techniques, Meditation)
Started | 100
Completed | 88
Not Completed | 12
Not completed — Time constraints | 2
Not completed — Health issues | 1
Not completed — Death in the family | 1
Not completed — Disliked the intervention | 1
Not completed — No reasons specified | 7

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (Video, Breathing Techniques, Meditation)
Number analyzed (Participants) | 100
Age, Customized [Count of Participants; unit: Participants]
  26-35 years | 33
  36-45 years | 22
  46-55 years | 25
  56-65 years | 18
  Above 66 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 72
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 19
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 60
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 100
Education [Count of Participants; unit: Participants]
  Junior/High | 9
  College | 20
  Masters or higher | 71
Religion [Count of Participants; unit: Participants]
  Catholic | 32
  Protestant | 33
  None | 20
  Other | 15
Occupation [Count of Participants; unit: Participants]
  Clinical role | 28
  Administration | 38
  Research | 27
  Unknown | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Recruited to the Study (Feasibility)
Description: To demonstrate the feasibility of a short pranayama or breathing techniques and meditation during Covid-19 pandemic. Feasibility will be defined as recruitment of 50 participants to the study within 2 months.
Time Frame: Within 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Video, Breathing Techniques, Meditation)
Number analyzed (Participants) | 100
Participants | 100

2. Primary Outcome: Number of Participants Who Perceived the Intervention as Useful
Description: Defined as more than 50% of participants perceive the intervention as useful. Meditation perception questions were asked such as usefulness, feeling at peace, hopeful, or relaxed, and responses were recorded as strongly agree, agree, neutral, disagree, and strongly disagree at weeks 1 and 4.
Time Frame: Week 1 and Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Video, Breathing Techniques, Meditation)
Number analyzed (Participants) | 100
Participants
  Week 1 | 69
  Week 4 | 56

3. Secondary Outcome: Change in Resilience
Description: Measured by the Brief Resilient Coping Scale among health care workers questionnaire.
Time Frame: 4 weeks
Reporting Status: Not Posted, anticipated posting 2027-11

4. Secondary Outcome: Perceive Stress and Psychological Impact
Description: Measured by the Perceived Stress Scale and COVID-19 Stress among health care workers questionnaire.
Time Frame: 4 weeks
Reporting Status: Not Posted, anticipated posting 2027-11

5. Secondary Outcome: Breath Holding Time
Description: Will determine the differences in breath holding time between those who are adherent and those who are not adherent to the practice.
Time Frame: 4 weeks
Reporting Status: Not Posted, anticipated posting 2027-11

6. Secondary Outcome: Adherence to the Practice
Description: Will determine the adherence to the practice assessed as at least 50% of participants implement the intervention for 3 or more times in a week by the end of week 1/day 7 (+ 3 days).
Time Frame: 4 weeks
Reporting Status: Not Posted, anticipated posting 2027-11

ADVERSE EVENTS:
Time Frame: adverse event data were collected at week 1 and week 4
Arm/Group | Supportive Care (Video, Breathing Techniques, Meditation)
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

LIMITATIONS AND CAVEATS:
Reporting Results for Primary Outcome Measures due to the PCD has been met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT04482647/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT04482647/ICF_001.pdf